CLINICAL TRIAL: NCT04114162
Title: Body Composition Monitor to Quantify Fluid Overload Related to Vascular Leak in Septic Shock Patients
Brief Title: Fluid Overload Quantification in Septic Shock
Acronym: FOTOShock
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Collaborators: Don du Souffle de Besançon (Unknown); Hopital Lariboisière (Other)
Responsible Party: Sponsor
Other Study IDs: P/2019/411
Record Dates: First submitted 2019-10-01; First posted 2019-10-03 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-01

CONDITIONS: Intensive Care Units; Shock, Septic
Keywords: ICU; Septic shock; Fluid overload; Quantification; Bioimpedancemetry; Capillary leak; Fluid responsiveness
MeSH Terms: conditions — Shock, Septic; Edema

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Fluid management in septic shock patients remain a great challenge. Insufficient fluid filling lead to hypovolemia, organ failure and increased death, whereas fluid overload was associated to an increased morbidity and mortality in several studies.

Several invasive and non invasive strategies have been developed during the past years to monitor the hemodynamic state of septic shock patients, but no method has been validated to objectively quantify fluid overload in septic shock patients.

The Body Composition Monitor (BCM) allow for measurement of total body water (TBW), extracellular water (ECW) and intracellular water (ICW) volumes using bioimpedancemetry. The BCW is daily used in patients who undergo renal dialysis to assess the effectiveness of fluid removal. The BCM has never been validated in septic shock patients.

The aim of the study is to investigate the accuracy of the BCM to measure the variation of the TBW during a fluid challenge of 500 ml of saline during the early phase of septic shock.

DETAILED DESCRIPTION:
Patients suffering from septic shock admitted in our critical care unit for less than 24 hours will be eligible. TBW, ECW and ICW volumes will be measured using the BCM just before (T0), just at the end (T1) and 1 h after the end (T2) of a fluid challenge of 500 ml of saline. Fluid responsiveness will be assessed using trans thoracic echocardiography (TTE). TTE will be performed at T0, T1 and T2. Blood samples will be obtained at T0, T1 and T2 to dose biomarkers of endothelial dysfunction and of capillary leak. The effectiveness of fluid challenge on microcirculation will be investigated by measuring the tissue perfusion index of the urethral mucosa using the IKORUS UP device.

Patients will be followed until Day 28 after admission in the critical care unit.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged from 18 to 80 years old
* Admitted to ICU for septic shock for less than 24 h
* Fluid resuscitation decided by intensivist
* Patient affiliated to a social security system or recipient of a such system
* Patient/proxy not opposed to the study

Exclusion Criteria:

* Subject with amputation of 1 or more limbs
* Body mass index > 35 kg.m-2 ou < 18 kg.m-2
* Impossibility of setting up an arterial catheter for invasive blood pressure monitoring and / or a central venous catheter in the upper cava territory
* Patient with pacemaker and / or implantable cardioverter defibrillator
* Quality of cardio echo image insufficient to allow studied parameters measurement
* Moribund subject ( life expectancy expected less than 48 hours)
* Uncontrolled intracranial hypertension (intracranial pressure ≥ 20 mm Hg by ICP monitoring or by a pulsatility index ≥ 1.30 in the transcranial Doppler)
* Patient under ECMO/ECLS
* Legal incapacity or limited legal capacity
* Subject without health insurance
* Pregnant woman
* Subject being in the exclusion period of another study or provided for by the "National Volunteer File"

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ICU patient requiring fluid resuscitation for septic shock
Sampling Method: Non-Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
To assess the accuracy of the BCM to measure the variation of the TBW volume during a fluid challenge. | 10 minutes
  The variation of the TBW volume measured by the BCM will be compared to the variation of the volume of fluids (fluid input minus fluid output) during a fluid challenge of 500 ml of saline. Fluid input will be the sum of the volume of all fluids and drugs delivered during the fluid challenge (including enteral nutrition). Fluid output will be the sum of all loss of fluid (surgical drain, urine output) during the fluid challenge.

SECONDARY OUTCOMES:
To describe the variation of the ECW volume measured by the BCM during a fluid challenge of 500 ml of saline. | 10 minutes
  The variation of the ECW volume during a fluid challenge of 500 ml of saline will be the difference between the ECW volume measured à T0 (just before the fluid challenge) and the ECW volume measured at T1 (just after the end of the fluid challenge).
To describe the variation of the ECW volume on TBW volume ratio during a fluid challenge of 500 ml of saline. | 10 minutes
  ECW and TBW volumes will be measured using the BCM just before the fluid challenge (T0) and just after the end of the fluid challenge (T1). The ECW volume on TBW volume ratio (ECW/TBW ratio) will be calculated at T0 and at T1. The variation of the ECW/TBW ration will be the difference between the ECW/TBW ratio measured at T0 and the ECW/TBW ratio measured at T1.
To compare the phase angle value measured at T0 by the BCM between responders and non responders at T1. | 10 minutes
  Fluid responsiveness at T1 will be defined by an increased of the stroke volume > 10% between T0 and T1. Stroke volume will be measured using trans thoracic echocardiography. The phase angle value at T0 will be compared between responders (patients with an increase of the stroke volume > 10%) and non responders.
To describe the relationship between the phase angle value measured at T0 by the BCM and the capillary leak index. | 10 minutes
  The capillary leak index is defined by the following ratio: (blood C-reactive protein*100)/(blood albumin).
To compare the ECW/TBW ratio at T0 between responders and non responders at T1. | 10 minutes
To compare the TBW volume at T0 between responders and non responders at T2. | 70 minutes
  Fluid responsiveness will be assessed at T2 (1 h after the end of the fluid challenge) using transthoracic echocardiography (TTE). Fluid responsiveness at T2 will be defined by an increased of the stroke volume > 10% compared to baseline (T0).
To compare the ECW/TBW ratio at T0 between responders and non responders at T2. | 70 minutes
  Fluid responsiveness will be assessed at T2 (1 h after the end of the fluid challenge) using transthoracic echocardiography (TTE). Fluid responsiveness at T2 will be defined by an increased of the stroke volume > 10% compared to baseline (T0).
To compare the ECW/TBW ratio at T2 between responders and non responders at T2. | 70 minutes
  Fluid responsiveness will be assessed at T2 (1 h after the end of the fluid challenge) using transthoracic echocardiography (TTE). Fluid responsiveness at T2 will be defined by an increased of the stroke volume > 10% compared to baseline (T0). ECW/TBW ratio will be calculated at T2 from the ECW and TBW volumes measured using the BCM at T2 (1 h after the end of fluid challenge).
To describe the variation of the tissue perfusion index of the urethral mucosa (uPI) measured using the IKORUS UP device during the fluid challenge of 500 ml of saline. | 70 minutes
  The uPI will be continuously measured during the fluid challenge and until 1 hours after the end of the fluid challenge. The uPI will be measured using the IKORUS UP device.
To describe the relationship between blood biomarkers of endothelial dysfunction and fluid responsiveness. | 70 min
  Blood biomarkers of endothelial dysfunction will be measured from blood samples obtained at T0, T1 and T2. Fluid responsiveness will be assessed using TTE. Fluid responsiveness will be defined by an increased of the stroke volume > 10% compared to baseline (T0).
To describe the relationship between blood biomarkers of capillary leak and fluid responsiveness. | 70 minutes
  Blood biomarkers of capillary leak will be measured from blood samples obtained at T0, T1 and T2. Fluid responsiveness will be assessed using TTE. Fluid responsiveness will be defined by an increased of the stroke volume > 10% compared to baseline (T0).

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Universitaire de Besançon, Besançon, France